CLINICAL TRIAL: NCT02986139
Title: A Multicenter, Randomized, Double-blind, Crossover Study to Assess the Injection Site Pain Associated With a Modified Etanercept Formulation in Adult Subjects With Either Rheumatoid Arthritis or Psoriatic Arthritis
Brief Title: Study to Assess the Injection Site Pain Associated With a New Etanercept Formulation in Adults With Rheumatoid Arthritis or Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20140339
Record Dates: First submitted 2016-11-02; First posted 2016-12-08 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Arthritis, Rheumatoid; Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence AB (Experimental): Participants received a single 50 mg subcutaneous (SC) dose of the commercial formulation etanercept in a prefilled SureClick autoinjector on day 1 (Treatment A) followed by a single 50 mg SC dose of the new formulation of etanercept in a prefilled SureClick autoinjector on day 8 (Treatment B).
  Interventions: Drug: Commercial Formulation Etanercept; Drug: New Formulation Etanercept
- Sequence BA (Experimental): Participants received a single 50 mg SC dose of the new formulation of etanercept in a prefilled SureClick autoinjector on day 1 (Treatment B) followed by a single 50 mg SC dose of the commercial formulation etanercept in a prefilled SureClick autoinjector on day 8 (Treatment A).
  Interventions: Drug: Commercial Formulation Etanercept; Drug: New Formulation Etanercept

INTERVENTIONS:
Drug: Commercial Formulation Etanercept — Etanercept was supplied in a single-use SureClick autoinjector as a sterile, preservative-free solution for SC injection containing 0.98 mL of 50 mg/mL etanercept in the commercial formulation.
  Other Names: Enbrel
Drug: New Formulation Etanercept — Etanercept was supplied in a single-use SureClick autoinjector as a sterile, preservative-free solution for SC injection containing 0.98 mL of 50 mg/mL etanercept in the new formulation.

SUMMARY:
The primary objective was to assess the injection site pain associated with the new formulation of etanercept compared with commercial etanercept in adults with rheumatoid arthritis (RA) or psoriatic arthritis (PsA) as measured by a visual analog scale (VAS).

DETAILED DESCRIPTION:
This is a phase 3b, multicenter, randomized, double-blind, 2-period, 2-sequence crossover study in adults with RA or PsA who are naive to etanercept. The study will evaluate injection site pain associated with the commercial formulation of etanercept and the new formulation of etanercept immediately after injection of each formulation.The study will consist of a screening period of up to 14 days, a 2 week treatment period with a 30 day post treatment safety follow-up. Each dose will follow the recommended label dosing for adults with RA and PsA: 50 mg weekly (scheduled approximately 7 days apart).

ELIGIBILITY:
Inclusion Criteria

* Subject has provided informed consent prior to initiation of any study specific activities/procedures.
* Male or female subject is 18 years of age or older at time of signing the informed consent form.
* Subject has a diagnosis of RA or PsA and indicated for treatment with etanercept per the current label, based on investigator judgment.
* Subject is naïve to etanercept.
* Subject is able to self-inject etanercept.

Exclusion Criteria

* Subject is diagnosed with Felty's syndrome.
* Subject has active erythrodermic, pustular, guttate psoriasis, or medication induced psoriasis, or other skin conditions.
* Subject has a history of clinically significant skin allergies
* Subject has a history of alcoholic hepatitis, nonalcoholic steatohepatitis or immunodeficiency syndromes.
* Subject has any active infection for which anti-infectives were indicated within 4 weeks prior to screening.
* Subject has had a serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to first dose of investigational product.
* Subject had prosthetic joint infection within 5 years of screening or native joint infection within 1 year of screening.
* Subject has known alcohol addiction or dependency.
* Subject has positive hepatitis B surface antigen, hepatitis B core antibody (confirmed by hepatitis B virus deoxyribonucleic acid (DNA) test) or hepatitis C virus antibody serology at screening, or a positive medical history for hepatitis B or C. (Subjects with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll).
* Subject has any active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma.
* Subject has known history of active tuberculosis.
* Subject has used biologic disease modifying agent (DMARD) less than or equal to 3 months prior to screening.
* If subject is receiving continuous treatment with acetaminophen, non-steroidal anti-inflammatory drug or tramadol, hydrocodone, oxycodone, codeine, and/or propoxyphene and the dose is within 4 hours before study visit and dose is not stable for ≥ 2 weeks before first dose of investigational product
* For subjects not on continuous analgesics, subject has taken the following within 4 hours before screening: acetaminophen, non-steroidal anti-inflammatory drugs, hydrocodone, codeine, tramadol, propoxyphene, and/or oxycodone (unless in the form of OxyContin). For subjects not on continuous analgesics, subject has taken OxyContin within 24 hours before screening.
* Subject has received live vaccines less than or equal to 4 weeks prior to first dose of investigational product.
* Subject has laboratory abnormalities during screening.
* Estimated creatinine clearance less than 50 mL/min.
* Subject has any other laboratory abnormality, which, in the opinion of the investigator poses a safety risk, will prevent the subject from completing the study, or will interfere with the interpretation of the study results.
* Subject is currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s).
* Other investigational procedures while participating in this study.
* Women who are pregnant or breastfeeding, or planning to become pregnant or breastfeed during treatment and/or within 4 weeks after the last dose of etanercept.
* Women of child-bearing potential with a positive pregnancy test.
* Women of child-bearing potential who are unwilling to practice true sexual abstinence or unwilling to use 1 of the following effective birth control methods during treatment and for an additional 4 weeks after the last dose of etanercept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (29):
  - Research Site, Birmingham, Alabama
  - Research Site, El Cajon, California
  - Research Site, Lomita, California
  - Research Site, Sherman Oaks, California
  - Research Site, Thousand Oaks, California
  - Research Site, Cutler Bay, Florida
  - Research Site, DeLand, Florida
  - Research Site, Doral, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Quincy, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Bay City, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Freehold, New Jersey
  - Research Site, Smithtown, New York
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, The Woodlands, Texas
  - Research Site, Bothell, Washington
  - Research Site, South Charleston, West Virginia
- Research Site, Ponce, Puerto Rico

REFERENCES:
- [Background] Cohen S, Samad A, Karis E, Stolshek BS, Trivedi M, Zhang H, Aras GA, Kricorian G, Chung JB. Decreased Injection Site Pain Associated with Phosphate-Free Etanercept Formulation in Rheumatoid Arthritis or Psoriatic Arthritis Patients: A Randomized Controlled Trial. Rheumatol Ther. 2019 Jun;6(2):245-254. doi: 10.1007/s40744-019-0152-8. Epub 2019 Mar 27. PMID 30915626
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 23 centers in the United States. The first participant enrolled on 29 November 2016 and the last participant enrolled on 01 September 2017.
Pre-assignment Details: Participants were randomized 1:1 to receive each etanercept formulation in 1 of 2 treatment sequences: AB (treatment A followed by treatment B) or BA (treatment B followed by treatment A).
Period: Overall Study
Arm/Group | Sequence AB | Sequence BA
Started | 56 | 55
Received Etanercept | 56 | 53
Completed | 55 | 51
Not Completed | 1 | 4
Not completed — Sponsor Decision | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence AB | Sequence BA | Total
Number analyzed (Participants) | 56 | 55 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (13.9) | 55.9 (13.7) | 55.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 41 | 77
  Male | 20 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 14 | 42
  Not Hispanic or Latino | 28 | 41 | 69
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Black or African American | 5 | 3 | 8
  Multiple | 1 | 0 | 1
  White | 50 | 50 | 100
Actual Indication [Count of Participants; unit: Participants]
  Rheumatoid Arthritis | 41 | 45 | 86
  Psoriatic Arthritis | 15 | 10 | 25

OUTCOME MEASURES:

1. Primary Outcome: Injection Site Pain
Description: Injection site pain was assessed using a 100 mm visual analog scale (VAS), from 0 mm (No Pain At All) to 100 mm (Worst Pain Imaginable). Participants were asked to indicate the severity of their pain at the injection site by placing a vertical line on the scale.
Time Frame: Immediately following injection of each study drug on day 1 and day 8 of this crossover study
Population: The primary analysis set included all participants who received both doses of commercial and new etanercept during each study period and who completed the injection site pain score during both study periods.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Etanercept Commercial Formulation: Participants received a single 50 mg SC dose of etanercept commercial formulation on either day 1 or day 8.
- Etanercept New Formulation: Participants received a single 50 mg SC dose of etanercept new formulation on either day 1 or day 8.
Arm/Group | Etanercept Commercial Formulation | Etanercept New Formulation
Number analyzed (Participants) | 104 | 104
mm | 23.6 (22.3) | 19.8 (22.5)
Statistical Analysis 1: Comparison: Etanercept Commercial Formulation vs Etanercept New Formulation; A mixed effects analysis of variance model was used to assess injection site pain with the new formulation of etanercept as the test treatment and the commercial formulation of etanercept as the reference treatment. Treatment, study period, sequence, and disease indication were evaluated as fixed effect covariates, and subject within sequence was included as a random effect; Test type: Superiority; p = 0.048, Mixed effects analysis of variance model; LS Mean Difference = -4.0, 95% CI 2-sided [-8.0 to -0.0]

2. Secondary Outcome: Injection Site Pain by Disease Indication
Description: as for outcome 1
Time Frame: Immediately following injection of each study drug on day 1 and day 8 of this crossover study
Population: Primary analysis set
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Etanercept Commercial Formulation - RA: Participants with rheumatoid arthritis (RA) received a single 50 mg SC dose of etanercept commercial formulation.
- Etanercept Commercial Formulation - PsA: Participants with psoriatic arthritis (PsA) received a single 50 mg SC dose of etanercept commercial formulation.
- Etanercept New Formulation - RA: Participants with RA received a single 50 mg SC dose of etanercept new formulation.
- Etanercept New Formulation - PsA: Participants with psoriatic arthritis (PsA) received a single 50 mg SC dose of etanercept new formulation.
Arm/Group | Etanercept Commercial Formulation - RA | Etanercept Commercial Formulation - PsA | Etanercept New Formulation - RA | Etanercept New Formulation - PsA
Number analyzed (Participants) | 81 | 23 | 81 | 23
mm | 23.7 (20.2) | 23.3 (29.0) | 20.5 (22.6) | 17.2 (22.3)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event was graded by the investigator using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: From first dose of etanercept to 30 days after the last dose; 38 days.
Population: The safety analysis set included all participants who received at least 1 dose of etanercept during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept Commercial Formulation | Etanercept New Formulation
Number analyzed (Participants) | 106 | 107
Participants
  All adverse events | 10 | 8
  Serious adverse events | 0 | 1
  AE leading to discontinuation of etanercept | 1 | 3
  Fatal adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of etanercept to 30 days after the last dose; 38 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Etanercept Commercial Formulation | Etanercept New Formulation
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/107
Serious Adverse Events (participants affected / at risk) | 0/106 | 1/107
Other Adverse Events (participants affected / at risk) | 10/106 | 7/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Commercial Formulation (N=106) | Etanercept New Formulation (N=107)
Bronchitis viral (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Commercial Formulation (N=106) | Etanercept New Formulation (N=107)
Nausea (Gastrointestinal disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 1
Injection site papule (General disorders) | 0 | 1
Injection site reaction (General disorders) | 2 | 1
Injection site swelling (General disorders) | 1 | 0
Injection site warmth (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Limb operation (Surgical and medical procedures) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02986139/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/39/NCT02986139/SAP_001.pdf